CLINICAL TRIAL: NCT01944293
Title: Ketamine vs. Midazolam in Bipolar Depression
Brief Title: Ketamine for Suicidality in Bipolar Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Michael Grunebaum, MD, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #6785
Record Dates: First submitted 2013-09-08; First posted 2013-09-17 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Bipolar Disorder; Major Depressive Episode; Suicidal Ideation
Keywords: Ketamine; Midazolam; Bipolar Disorder; Major Depressive Episode; Suicidal Ideation; Suicide; Depression; Treatment; Ketamine Treatment
MeSH Terms: conditions — Bipolar Disorder; Suicidal Ideation; Suicide; Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): 0.5 mg/kg, I.V. (in the vein)
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): 0.02 mg/kg, I.V. (in the vein)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — Single dose of 0.5 mg/kg of Ketamine given intravenously (in the vein) over 40 minutes
  Other Names: Ketalar; Ketamine Hydrochloride Injection
  Arms: Ketamine
Drug: Midazolam — Single dose of 0.02 mg/kg of Midazolam given intravenously (in the vein) over 40 minutes
  Other Names: Midazolam Injection
  Arms: Midazolam

SUMMARY:
This study is designed to compare the effectiveness of two medications, Ketamine and Midazolam, for rapidly relieving suicidal thoughts in people suffering from bipolar depression.

The first drug, ketamine, is an experimental antidepressant that early studies have shown may quickly reduce suicidal thoughts, but we are not sure how well it may work. Midazolam, the comparison drug, is not thought to reduce depression or suicidal thoughts.

DETAILED DESCRIPTION:
Patients currently taking psychiatric medications may continue them during the study. However, if a patient is taking a benzodiazepine (such as Ativan, Klonopin, or Xanax), they will be able to take up to 2mg per day of Lorazepam during the week before the infusion, but none will be permitted in the 24 hours pre-infusion. Also, Zolpidem (Ambien) will not be permitted in the 24 hours pre-infusion. If a person chooses to participate, their dose of benzodiazepine may need to be reduced so that they can do without it during the 24 hours pre-infusion.

Participants are randomly assigned to receive a single dose of Ketamine (0.5 mg/kg) or Midazolam (0.02 mg/kg), which is given slowly, in a vein, over about 40 minutes. The study is "double-blind," meaning patients and study staff will not know which medication is in the infusion.

If a patient does not respond to the first infusion, and s/he received Midazolam, then s/he will be offered the option of a second infusion, this time with Ketamine (0.5 mg/kg). After the infusion(s), participants will have weekly research interviews for 6 weeks to monitor response.

After post-infusion research measures are completed, all subjects will receive open clinical treatment. During open clinical treatment, medication will be changed for those patients who don't respond or whose response is transient.

Participation in this study requires a brief inpatient stay, at no cost, at the New York State Psychiatric Institute (NYSPI).

Eligible participants enrolled in this study will be offered medication management visits at no cost for a total of up to 6 months combining inpatient and outpatient treatment. At the end of the 6 months of treatment patients will be referred for ongoing care.

ELIGIBILITY:
INCLUSION CRITERIA:

* Bipolar depression with current major depressive episode (MDE). Participants may be psychiatric medication-free, or if on psychiatric medication, not responding adequately given current MDE with suicidal ideation.
* Moderate to severe suicidal ideation
* 18-65 years old
* Patients will only be enrolled if they agree to voluntary admission to an inpatient research unit at the New York State Psychiatric Institute (NYSPI) for infusion phase of treatment.
* Pre-menopausal female participants of child-bearing potential must be willing to use an acceptable form of birth control during study participation such as condoms, diaphragm, oral contraceptive pills
* Able to provide informed consent
* Subjects 61-65 years old must score 25 or higher on the Mini-Mental State Examination (MMSE) at screening

EXCLUSION CRITERIA:

* Unstable medical condition or neurological illness, including baseline hypertension (BP>140/90) or significant history of cardiovascular illness
* Significant ECG abnormality
* Pregnancy and/or lactation
* Current psychotic symptoms
* Contraindication to any study treatment
* Current or past ketamine abuse or dependence ever (lifetime); any other drug or alcohol dependence within past 6 months; suicidality only due to binge substance use or withdrawal
* Inadequate understanding of English
* Prior ineffective trial of or adverse reaction to ketamine or midazolam
* Opiate use greater than total daily dose of 20mg Oxycodone or equivalent during the 3 days pre-infusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-09; Primary Completion 2017-09 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Grunebaum, M.D., Principal Investigator — Columbia Unviversity/New York State Psychiatric Institute
Locations (1):
- Columbia University/New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: MIND Clinic for Mood and Personality Disorders — http://www.columbiapsychiatry.org/mind/

RESULTS

PARTICIPANT FLOW:
Groups:
- Midazolam: 0.02 mg/kg, I.V. (in the vein)
  Ketamine: Single dose of 0.5 mg/kg of Ketamine given intravenously (in the vein) over 40 minutes
  Midazolam: Single dose of 0.02 mg/kg of Midazolam given intravenously (in the vein) over 40 minutes
Period: Overall Study
Arm/Group | Ketamine | Midazolam
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Midazolam | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (10.2) | 43 (13.9) | 40.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity, Customized: Non-white
  Participants
    More than one race | 1 | 0 | 1
    White race | 6 | 8 | 14
    Not Hispanic | 7 | 8 | 15
    Hispanic | 0 | 1 | 1
    Asian | 0 | 1 | 1
Beck Scale for Suicidal Ideation (Clinician-rated) [Mean (Standard Deviation); unit: units on a scale] — This scale has 19 items scaled 0 (least severe) to 2 (most severe) with a potential score total range of 0 to 38 measuring severity of suicidal thoughts.
  units on a scale | 16.7 (8.4) | 16.8 (6.0) | 16.8 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Suicidal Ideation Measured With the Beck Scale for Suicidal Ideation
Description: Change in suicidal ideation in Bipolar Disorder during a Major Depressive Episode (MDE), with moderate to severe suicidal thoughts, from the pre-infusion baseline to 24 hours after the infusion of Ketamine (study drug) or Midazolam (active control).
Time Frame: At 24 hours post-Infusion
Population: Bipolar depression with suicidal ideation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 7 | 9
units on a scale | -12.4 (11.6) | -6.7 (7.4)

2. Secondary Outcome: Change in Systolic Blood Pressure
Description: Blood pressure is measured in millimeters of mercury.
Time Frame: During study infusion
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Ketamine | Midazolam
Number analyzed (Participants) | 7 | 9
mm Hg | 23 (12.8) | 3 (10.2)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ketamine | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 4/7 | 0/9
Other Adverse Events (participants affected / at risk) | 0/7 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=7) | Midazolam (N=9)
Increased suicidal thoughts requiring hospitalization (Psychiatric disorders) | 2 (4) | 0 (0)
suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Preparatory suicidal behavior (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT01944293/SAP_001.pdf
  • Study Protocol (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT01944293/Prot_002.pdf